CLINICAL TRIAL: NCT06781619
Title: Effect of Plant Based High Energy High Protein Oral Nutritional Supplement on Nutritional Intake in Patients With or at Risk of Disease Related Malnutrition.
Acronym: PRO-PLANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 23REX0061267
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Disease Related Malnutrition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant Based High Energy High Protein (PB HEHP) Oral Nutrition Supplement (ONS) (Experimental): Test Product
  Interventions: Dietary Supplement: Test Product: Plant based high energy high protein ONS
- Diary Based High Energy High Protein (DB HEHP) Oral Nutrition Supplement (ONS) (Active Comparator): Control Product
  Interventions: Dietary Supplement: Control Product: Dairy based high energy high protein ONS

INTERVENTIONS:
Dietary Supplement: Test Product: Plant based high energy high protein ONS — Plant based high energy high protein ONS 2 servings/day for a period of 8 weeks.
  Arms: Plant Based High Energy High Protein (PB HEHP) Oral Nutrition Supplement (ONS)
Dietary Supplement: Control Product: Dairy based high energy high protein ONS — Dairy based high energy high protein ONS 2 servings equivalent in energy & protein for a period of 8 weeks.
  Arms: Diary Based High Energy High Protein (DB HEHP) Oral Nutrition Supplement (ONS)

SUMMARY:
The subjects will use study product twice daily for 8 weeks starting at Visit 1. The recommendation is to consume one serving in the morning and one in the afternoon / evening between meals. The duration of the study for each subject will be approximately 11 weeks, comprising a screening period of max 2 weeks, an intervention period of 8 weeks, and a follow up phone call 1 week after completion of the intervention. A blood sample will be drawn at visit 1 and visit 3.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Identified as at medium or high risk of malnutrition based on:

   1. MUST score ≥ 1 and / or
   2. Being prescribed with ONS and willing and able to switch from pre-study prescribed ONS to the Test or Control Product for participation in the study
3. In need of 2 servings of ONS/day (400 kcal; 20 gr protein per serving) for at least 8 weeks as determined by the treating healthcare professional.
4. Medically and physically able to consume high energy high protein ONS in the opinion of the Investigator.
5. Willing to maintain dietary habits for the duration of the study.
6. Willing to consume plant based as well as dairy based ONS

Exclusion Criteria:

1. Known allergy to soy, cow's milk protein or to any other ingredients as listed in the study product composition (refer to the product information brochure (PIB) and the appendix of this protocol).
2. Known intolerance to any ingredients as listed in the study product composition (refer to PIB and appendix of this protocol). Subjects with lactose intolerance who use lactase may still be enrolled in the study.
3. Any contraindication to oral feeding per se, including gastrointestinal failure or suppressed gastrointestinal function, complete intestinal obstruction and major intraabdominal sepsis.
4. Active flare of inflammatory bowel disease as defined by Harvey-Bradshaw Index (HBI) >6 (Crohn's disease) or Simple Clinical Colitis Activity Index (SCCAI) >5 (ulcerative colitis).
5. Requiring a protein restricted diet as confirmed by a physician, for example chronic kidney disease stage 4 and 5 (estimated by Glomerular Filtration Rate <30 mL/min/1.73 m2).
6. Requiring enteral nutrition (via tube delivery) or parenteral nutrition.
7. Subjects following a vegan diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To investigate the effect of PB HEHP ONS compared to DB HEHP ONS on nutritional intake (energy & protein) in subjects with or at risk of Disease Related Malnutrition (DRM) and/or prescribed with ONS. | 11 weeks
  Mean total protein intake and mean total energy intake in subject with or at risk of Disease Related malnutrition (DRM) and/or prescribed with ONS will be measured by 3-day nutritional intake diary at baseline, at week 4 and week 8.

CONTACTS AND LOCATIONS:
Locations (2):
- Meclinas, Mechelen, Belgium
- QClinical, Rotterdam, Netherlands